CLINICAL TRIAL: NCT06208423
Title: Management Reasoning With AI Chat Bots
Brief Title: Physician Reasoning on Management Cases With Large Language Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Jonathan Chen, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71319b
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Clinical Decision-making
Keywords: clinical decision support

STUDY DESIGN:
Intervention Model Description: The trial will be designed as a randomized, two-arm, single-blind parallel group study.
Who Masked: Outcomes Assessor
Masking Description: The grading of responses will be performed by assessors blinded to participant identity and treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPT-4 (Active Comparator): Group will be given access to GPT-4
  Interventions: Other: GPT-4
- Usual Resources (No Intervention): Group will not be given access to GPT-4 but will be encouraged to use any resources they wish besides large language models (UpToDate, Dynamed, google, etc).

INTERVENTIONS:
Other: GPT-4 — OpenAI's GPT-4 large language model with chat interface.
  Arms: GPT-4

SUMMARY:
This study will evaluate the effect of providing access to GPT-4, a large language model, compared to traditional management decision support tools on performance on case-based management reasoning tasks.

DETAILED DESCRIPTION:
Artificial intelligence (AI) technologies, specifically advanced large language models like OpenAI's ChatGPT, have the potential to improve medical decision-making. Although ChatGPT-4 was not developed for its use in medical-specific applications, it has demonstrated promise in various healthcare contexts, including medical note-writing, addressing patient inquiries, and facilitating medical consultation. However, little is known about how ChatGPT augments the clinical reasoning abilities of clinicians.

Clinical reasoning is a complex process involving pattern recognition, knowledge application, and probabilistic reasoning. Integrating AI tools like ChatGPT-4 into physician workflows could potentially help reduce clinician workload and decrease the likelihood of mismanagement. However, ChatGPT-4 was not developed for clinical reasoning nor has it been validated for this purpose. Further, it may be subject to disinformation, including convincing confabulations that may mislead clinicians. If clinicians misuse this tool, it may not improve reasoning and could even cause harm. Therefore, it is important to study how clinicians use large language models to augment clinical reasoning prior to routine incorporation into patient care.

In this study, participants will be randomized to answer clinical management cases with or without access to ChatGPT-4. Each case has multiple components, and the participants will be asked to discuss their reasoning for each component. Answers will be graded by independent reviewers blinded to treatment assignment. A grading rubric was developed for each case by a panel of 4-7 expert discussants. Discussants independently developed a rubric for each case, and then any discrepancies were resolved through multiple rounds of discussions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be licensed physicians and have completed at least post-graduate year 2 (PGY2) of medical training.
* Training in Internal medicine, family medicine, or emergency medicine.

Exclusion Criteria:

* Not currently practicing clinically.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Management Reasoning | Within one-hour study
  Percent correct (range: 0 to 100) for each case.

SECONDARY OUTCOMES:
Time Spent on Management | Within one-hour study
  Time (in minutes) participants spend per case between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan H Chen, MD, PhD, Principal Investigator — Stanford University; Adam Rodman, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Andrew Olson, MD, Principal Investigator — University of Minnesota
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh E, Gallo RJ, Strong E, Weng Y, Kerman H, Freed JA, Cool JA, Kanjee Z, Lane KP, Parsons AS, Ahuja N, Horvitz E, Yang D, Milstein A, Olson APJ, Hom J, Chen JH, Rodman A. GPT-4 assistance for improvement of physician performance on patient care tasks: a randomized controlled trial. Nat Med. 2025 Apr;31(4):1233-1238. doi: 10.1038/s41591-024-03456-y. Epub 2025 Feb 5. PMID 39910272
- [Derived] Goh E, Gallo R, Strong E, Weng Y, Kerman H, Freed J, Cool JA, Kanjee Z, Lane KP, Parsons AS, Ahuja N, Horvitz E, Yang D, Milstein A, Olson APJ, Hom J, Chen JH, Rodman A. Large Language Model Influence on Management Reasoning: A Randomized Controlled Trial. medRxiv [Preprint]. 2024 Aug 7:2024.08.05.24311485. doi: 10.1101/2024.08.05.24311485. PMID 39148822